CLINICAL TRIAL: NCT03330522
Title: Reducing HIV Risk in Urban Women: Soap Opera Videos on Video-Capable Cell Phones
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northeastern University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: LSCR012008
Record Dates: First submitted 2017-10-23; First posted 2017-11-06 (Actual); Last update posted 2017-11-06 (Actual); Status verified 2017-10

CONDITIONS: HIV/AIDS; Sexual Behavior; Woman's Role; Risk Behavior
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Sexual Behavior; Risk-Taking | interventions — Sex

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): The active intervention is "Love, Sex, & Choices," a 12-episode, online HIV prevention intervention video series accessed on study provided smartphones. Each episode is up to 20 minutes in length. Study participants receive one episode per week for 12 weeks on study provided smartphones.
  Interventions: Other: Love, Sex, & Choices video series
- Control Comparison Group (Active Comparator): The control comparison intervention is twelve messages in text that promote HIV prevention behaviors and open communication with male sex partners. Study participants receive one message per week for 12 weeks on study provided smartphones.
  Interventions: Other: Messages in text

INTERVENTIONS:
Other: Love, Sex, & Choices video series — Love, Sex, and Choices was written and scripted by the study team and underwent pilot testing in the target population. The series was divided into 15-to-20 minute episodes that were streamed weekly. The principles of reducing HIV risk were communicated through the characters and high risk situations. The lead characters model how women become more powerful, meaning more aware of themselves as worthy of respect, making choices intentionally, feeling free to pursue their intentions, and involving themselves in creating change. This process leads to higher power sex scripts in the characters, meaning pursuing intentional choices and health promoting behaviors. The lead characters model open communication about HIV testing with a resistant partner, and initiating condom use.
  Arms: Intervention
Other: Messages in text — The comparison group received 12 weekly HIV health promotion written messages over the smartphone. The messages were based on prevailing CDC recommendations and the theoretical framework. An example is: "Sexual health means respecting your own rights and feelings. Feeling pressured to have sex means limiting your choices and your freedom to love safely. …. If he doesn't like you being you, it may be time to walk." Other messages provided instructions on the correct condom use and the importance of HIV testing. The 12 messages were reviewed by ten African American and Latina undergraduate nursing students for ease of comprehension.
  Arms: Control Comparison Group

SUMMARY:
Background: Love, Sex, and Choices (LSC) is a soap opera video series created to reduce HIV sex risk in women.

Methods: LSC was compared to text messages in a randomized trial in 238 high-risk mostly Black young urban women. 117 received 12-weekly LSC videos, 121 received 12-weekly HIV prevention messages on smartphones. Changes in unprotected sex with high risk partners were compared by mixed models.

DETAILED DESCRIPTION:
This randomized controlled trial (RCT) aims to evaluate "Love, Sex, & Choices" (LSC), a video-based intervention to reduce human immunodeficiency virus (HIV) sex risk behaviors in young adult urban women. Consisting of 12-weekly soap opera videos lasting up to 20 minutes each, messages about reducing HIV sexual risk are communicated through the drama and context of relationships, a strength of the soap opera modality. Based on true stories analyzed from focus groups, viewers can identify with the heroines in the videos who suffer tragedy and heartbreak and transform their behavior through a new awareness of their value as women, their choices, and their potential. Women watch a new video sequel weekly for 12 weeks on smartphones. A control group receives text/audio messages concerning HIV risk reduction. If successful, the public health impact is that women at risk for HIV will be able to access video interventions to reduce HIV risk on personal mobile devices.

Prior to this work, a 43-minute soap opera video, "A Story about Toni, Mike, and Valerie" had been produced and pilot tested by the Principal Investigator (PI) on handheld computers (RO3 NR009349). Findings had indicated the video was highly appealing and there was a statistically significant short-term reduction in stereotypical gender views about the need to engage in unprotected sex in the video intervention arm that was not observed in the control arm.

The current RCT seeks to test the effect of the LSC series on sex risk behavior as compared to a control receiving HIV prevention text messages. Analysis and story development had been guided by Sex Script Theory and the Theory of Power as Knowing Participation in Change; as well as, content analysis of focus groups with urban young adult African American and Latina women. Consistent with the theories and focus group analyses, the new LSC series elaborates on the original story weaving in the stories of four women. In both the RO3 pilot study and the related National Library of Medicine funded study (1 G08 LM008349-01), the use of small handheld computers to watch the video was found to be enjoyable and promoted a sense of privacy. Based on these promising findings concerning the experience of viewing videos on small handheld devices, the popularity of cell phones in this age group, and that the use of cell phones to watch videos is growing as cell phone technology, multimedia, and Internet connections improve, the present study seeks to deliver the weekly series of videos on smartphones.

There are several advantages of viewing videos on smartphones, in particular the freedom to watch the intervention videos often and in privacy. This study is also consistent with several NINR objectives stated in its strategic plan. These are: to apply findings concerning the social and cultural context of health behavior to health promotion, to develop and test interactive web-based and wireless technologies to eliminate health disparities, and to refine methods in the delivery of health promotion. The overall aim of this study is to conduct a RCT to determine whether the 12-week series of theory-based urban soap operas will reduce HIV sexual risk behavior. The specific aims of this study are:

Aim1. Complete final editing phase of LSC, a series of 12, 20-minute soap opera videos, and 12 HIV health promotion text/audio messages that will be released weekly and viewed on smartphones.

Aim 2. Deploy the web-based applications, specifically: a) integrate voice and text files into the audio computer assisted self-interview (ACASI) for access on desk top computers b) stream the videos to the video intervention group and send text/audio messages to the control group for viewing on smartphones c) maintain password protected availability so the video intervention group can watch the videos (or control group view text messages) anytime during the 12-weeks d) track how often and how long each video(or text) is viewed, and e) secure hardware and networks.

Aim 3. Conduct a RCT with 250 urban women aged 18 to 29 in two adjacent cities with a high incidence of HIV/AIDS. Inclusion criteria are women with high sex risk behavior. Eligibility screening will be accomplished by utilizing a previously developed ACASI that functions as a decision support system (DSS) to assign a level of risk based on responses to the screening interview. If supported by results, promote public access to the videos on the study dedicated web site.

The following hypotheses were tested in the RCT:

Primary hypotheses 1) The video group will have greater reductions in unprotected sex with all high risk sex partners (as measured by the USR score) from baseline to 3 and 6 months than will the control group. 2) The video group will have greater reduction in sexual pressure scores from baseline to 3 and 6 months than will the control group.

Secondary hypotheses: Compared to the control group, the video group will have 1) greater reductions in USR with high risk main partner/s from baseline to 3 and 6 months, 2) greater reductions in USR with non-main and secondary partners at 3 and 6 months, and, 3) The video group will have fewer high risk sex partners at 3 and 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Women 18-29 years old
* Unprotected vaginal or anal sex with at least one man that they perceive as engaging in risky behavior OR
* Unprotected vaginal or anal sex with more than 1 man regardless of perceived partner risk
* Can understand written and spoken English

Exclusion Criteria:

* Women younger than 18 years old
* Women older than 29 years old
* Cannot understand written or spoken English
* Previously participated in the study

Ages: 18 Years to 29 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Identify as female
Enrollment: 295 (Actual)
Dates: Start 2008-11-26 (Actual); Primary Completion 2011-03-16 (Actual); Study Completion 2014-02-28 (Actual)

PRIMARY OUTCOMES:
Change in unprotected sex risk with high risk partners from baseline to 6 months post-intervention | change in sex risk behavior from baseline to 6 months
  Sex risk is measured by the Vaginal Episode Equivalent (VEE) score (Susser, Desvarieux, & Wittkowski, 1998) with high risk partners. The VEE is the sum of all unprotected vaginal anal sex acts weighted by the relative HIV transmission risk (vaginal 1 and anal 2). A high risk partner is defined as the likelihood the male partner had sex with another woman, sex with men, or injected drugs in the past 3 months. Partner risk could range from 0 to 9; main or non-main partners with scores > 0 were considered to engage in risk behavior. Multiple partners were considered high-risk. An HIV positive partner is high risk.There is a four-point response metric, from "Definitely not" (0) to "Definitely did" (3). Only women having unprotected sex with a partner they perceived to have risk > 0 by this system were included into the study. For a given visit, unprotected vaginal and anal sex with all high risk partners in the previous 3 months were calculated at baseline and at 3 and 6 months.

CONTACTS AND LOCATIONS:
Overall Officials: Rachel Jones, PhD, Principal Investigator — Northeastern University
Locations (1):
- Northeastern University, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Jones R, Hoover DR, Lacroix LJ. A randomized controlled trial of soap opera videos streamed to smartphones to reduce risk of sexually transmitted human immunodeficiency virus (HIV) in young urban African American women. Nurs Outlook. 2013 Jul-Aug;61(4):205-215.e3. doi: 10.1016/j.outlook.2013.03.006. Epub 2013 Jun 4. PMID 23743482
- [Result] Jones R, Lacroix LJ. Streaming weekly soap opera video episodes to smartphones in a randomized controlled trial to reduce HIV risk in young urban African American/black women. AIDS Behav. 2012 Jul;16(5):1341-58. doi: 10.1007/s10461-012-0170-9. PMID 22430640
- See also: Link to main study publication — http://dx.doi.org/10.1016/j.outlook.2013.03.006